CLINICAL TRIAL: NCT03244852
Title: Patient-specific, Effective, and Rational Functional Connectivity Targeting for DBS in OCD
Acronym: PERFECT DBS
Status: Withdrawn | Type: Observational
Why Stopped: Data was analyzed from a previously collected dataset so no new participants were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Associate Professor of Psychiatry, Massachusetts General Hospital
Other Study IDs: 2017P000882
Record Dates: First submitted 2017-06-26; First posted 2017-08-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; deep brain stimulation; treatment-resistant OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OCD Patients with Deep Brain Stimulators: Patients with deep brain stimulation for intractable obsessive compulsive disorder (OCD)

SUMMARY:
The study aims to improve patient-specific anatomical targeting of the Deep Brain Stimulation for the treatment of intractable OCD.

DETAILED DESCRIPTION:
Recently, deep brain stimulation (DBS) has emerged as a potentially circuit-specific treatment for intractable OCD. DBS is programmable, allowing the clinician to "reshape" the volume of tissue activated within the standard ventral capsule/ventral striatum (VC/VS) target.

However, VC/VS DBS' efficacy is limited by two major factors: imperfect targeting and a lack of decision rules for stimulation adjustment. The VC/VS target is not a single identifiable structure, but encompasses white matter of the internal capsule and gray matter of the nucleus accumbens (NAc). In current practice for DBS in OCD, all patients are implanted at standard x,y,z coordinates in the VC/VS region. Due to this inter-subject anatomical variability, different fiber tracts are stimulated by ostensibly the "same" parameters in each subject, leading to variable outcomes. This investigation will identify aspects of VC/VS circuitry that may determine clinical response. The hypothesis is that good clinical outcomes may correlate to electrical field capture of either striatal gray matter or of white matter fibers connecting OFC to thalamus.

The current study looks to extend the neuroimaging investigation using anatomic white matter targeting, functional gray matter targeting and changes in changes in regional glucose metabolism of Deep Brain Stimulation (DBS) in severe obsessive-compulsive disorder (OCD) with the long-term aim of identifying biomarkers that could improve outcomes of this expensive and invasive therapy. Improved imaging would allow surgeons to place the DBS lead closer to the biological targets, thus improving efficacy of the treatment.

The objectives of this study are threefold:

* Improve the anatomic white matter targeting of the Deep Brain Stimulator (DBS) implant by tracing and identifying fibers of passage within the Ventral Capsule (VC) white matter using advance tractography methods in preoperative diffusion MRI data.
* Improve functional gray matter targeting by studying the overlap of the volume of tissue activated (VTA) with the VC voxels of maximal preoperative connectivity to the orbitofrontal cortex (OFC)
* Determine the changes in regional glucose metabolism using preoperative and post-treatment FDG-PET (Positron Emission Tomography) following 3 months of DBS treatment

ELIGIBILITY:
Inclusion Criteria:

1. OCD, diagnosed by Structured Clinical Interview for DSM-5 (SCID-5), judged of disabling severity with a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 28.
2. Persistence of severe symptoms and impairment for five or more years despite: i. at least three adequate (≥3 months at the maximum tolerated dose) serotonin transporter inhibitor trials (may use any serotonin or serotonin-norepinephrine inhibitors, but must include a trial of clomipramine) alone or in combination with ii. adequate behavior therapy (≥20 sessions of expert exposure and response prevention; At least 20 sessions of behavioral therapy must be attempted), and iii. augmentation of one of the selective SRIs with a neuroleptic or clonazepam.
3. Age between 21 and 64 years.
4. Able to understand and comply with instructions.
5. Able to give fully informed, written consent.
6. Approved to be implanted with a DBS device for OCD.

Exclusion Criteria:

1. Current or past psychotic disorder.
2. Full-scale IQ below 75 on the Wechsler Abbreviated Scale of Intelligence (WAIS) or cognitive impairment that would affect a participant's ability to give informed consent or provide interview or self-report data reliably, as determined by the consent monitor and the site psychiatrist. A questionnaire assessing consent comprehension will be used with all study subjects, to ensure that they understand the key procedures of the study, and its risks and benefits.
3. A clinical history of bipolar mood disorder; substance-induced mania is not an exclusion.
4. Any current clinically significant neurological disorder or medical illness affecting brain function, other than tic disorders or Tourette syndrome.
5. Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
6. Any labeled DBS contraindication, and/or inability to undergo presurgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation, significant cardiac or other medical risk factors for surgery.
7. Current or unstably remitted substance abuse, dependence, or a positive urine toxicology screen.
8. Pregnancy and women of childbearing age not using effective contraception.
9. Unable to adhere to operational and administrative study requirements (in the investigators' judgment).
10. Clinical history of severe personality disorder.
11. Imminent risk of suicide or an inability to control suicide attempts (in the investigators' judgment). History of serious suicidal behavior or one or more interrupted suicide attempts with potential lethality judged to result in serious injury or death.
12. Diagnosis of body dysmorphic disorder.
13. Evidence of dementia or other significant cognitive impairment on neuropsychological evaluation
14. Past or present diagnosis of hoarding disorder.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be 11 patients with DSM-5-defined OCD of disabling severity, refractory to prolonged treatment trials with conventional medication and behavioral therapy, who would therefore otherwise be candidates for psychiatric neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 6 months
  Yale-Brown Obsessive-Compulsive Scale (YBOCS) will be the principal outcome measure to correlate OCD symptoms severity.
Yale-Brown Obsessive-Compulsive Scale (YBOCS) and Neural Correlates (1) | 6 months
  Clinical improvement (change in YBOCS from baseline) will be correlated with the degree of postoperative capture of OFC fibers in the VTA of the active DBS contact
Yale-Brown Obsessive-Compulsive Scale (YBOCS) and Neural Correlates (2) | 6 months
  Clinical improvement (change in YBOCS from baseline) will be correlated with overlap of the volume of tissue activated (VTA) with the identified ventral striatum voxels of maximal preoperative connectivity to the OFC.
Yale-Brown Obsessive-Compulsive Scale (YBOCS) and Neural Correlates (3) | 6 months
  Clinical improvement (change in YBOCS from baseline) will be correlated with changes in regional glucose metabolism in the OFC, caudate, and thalamus.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No